CLINICAL TRIAL: NCT04734366
Title: Effect of the Baseball Suturing Technique on the Incidence of Isthmocele and Residual Myometrial Thickness After Cesarean: a Randomized Controlled Trial
Brief Title: Effect of Baseball Suturing on Isthmocele and Residual Myometrial Thickness After Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, İlhan Bahri Delibas, Tokat Gaziosmanpasa University, Head of Gynecology and Obstetrics Department, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GaziosmanpasaKHD
Record Dates: First submitted 2020-12-26; First posted 2021-02-02 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Isthmocele; Cesarean Section Complications
Keywords: isthmocele; baseball suture; cesarean

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uterine closure with "Baseball" suture technique (Experimental): Participants will undergo "Baseball" suture closure of the hysterotomy site at the time of cesarean section.
  Interventions: Procedure: Uterine closure with "Baseball" suture technique
- Single Layer Continuous Locked (Active Comparator): Participants will undergo Single Layer Continuous Locked suture closure of the hysterotomy site at the time of cesarean section.
  Interventions: Procedure: Single Layer Continuous Locked

INTERVENTIONS:
Procedure: Uterine closure with "Baseball" suture technique — A simple running (continuous) "baseball" suture is essentially an interrupted sutures. Applied as inside to outside/inside to outside of incision.
  Arms: Uterine closure with "Baseball" suture technique
Procedure: Single Layer Continuous Locked — Suturing is continued by passing through the previous stitch.
  Arms: Single Layer Continuous Locked

SUMMARY:
Cesarean delivery rates in Turkey as well as all over the world are increasing. Recent data in Turkey shows that the value of cesarean delivery rate reached 53%. This worldwide increase causes new concerns. Incomplete healing of the uterine scar after cesarean is a complication with potential long-term consequences. There is evidence that the risk of uterine scar defects is associated with the number of previous cesarean deliveries and the method of uterotomy closure. Study was designed as prospective randomized clinical trial to analyze the effects of two different uterine suture techniques. The investigators aim is to compare the closure of the incision with the "baseball" suture technique and the single-layer locking technique in terms of the incidence and depth of the isthmocele in the uterine incision scar as a short-term result.

DETAILED DESCRIPTION:
This study was designed as a double-blind randomized prospective and cross-sectional. Cesarean delivery planned patients who will admit to the Obstetrics and Gynecology Clinic, Tokat Gaziosmanpasa University Research and Application Center between January 2021 and June 2021 will be evaluated. Participation of the patients in the study will be based on written consents. All patients who meet the inclusion criteria will be randomized into two groups (i.e., "baseball" or single layer locked).

This study was approved by Tokat Gaziosmanpasa University Institutional Review Board and Ethics Committee (Project no= 20-KAEK-311, Approval Date= 12/17/2020).

Pregnant women who are over 37 weeks, have no pregnancy complications, and will undergo uterine surgery for the first time will be included in the study. Exclusion criteria are determined as: Preoperative hemogram value below 10mg/dL, active labor (regular contraction and> 4cm cervical opening), placental anomaly, previous uterine surgery, chorioamnionitis, premature rupture of membranes, additional disease, body mass index BMI> 35kg / m2, consuming tobacco and / or alcohol, needing blood transfusion and multiple pregnancy.

Randomization will be created on a computer controlled by a statistician to create two groups. Before cesarean delivery, sealed, opaque and numbered envelope containing the definition and image of the suture technique will be reported to the surgeon. Participants included in the study 3 months after the operation will be called for control by an external observer. Follow-up data and ultrasound measurements of uterine incision scar area will be documented by sonographer who does not know the uterotomy closure technique applied to the patient.

During the follow up examination, weight and breastfeeding status of the patient and ultrasound measurement of uterine length, uterine position, residual myometrial thickness, isthmocele depth, isthmocele width, cervical thickness, isthmocele fundus distance, isthmocele cervical distance, hypoechoic isthmocele width in transverse plane will be recorded.

The sample size was calculated based on a study by Roberge S et al. (2016) titled Impact of uterine closure on residual myometrial thickness after cesarean: a randomized controlled trial. The mean residual myometrial thickness values of this study were found to be 3.8 ± 1.57 in the single-layered group and 4.77 ± 1.34 in the double-stitched group. The power analysis performed using GPower 3.1 (http://www.gpower.hhu.de/) program, when 80% power and alpha = 0.05 are taken, the total sample size calculated using the student's t test was found to be 36 for each group. Considering possible problems, it is planned to include 80 participants, 40 for each group. The normal distribution of the data of the measurements will be analyzed with the Kolmogorov-Smirnov test. The data of two groups of patients will be analyzed with the Statistical Package for Social Sciences (SPSS) version 20 program using one-way ANOVA analysis, post-hoc test, T-test, chi-square and Fisher test according to the data characteristics. Statistical significance will be accepted as p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing their first cesarean section
* After 37 gestational week pregnancy
* Have no pregnancy complications

Exclusion Criteria:

* Preoperative hemogram value below 10mg / dl
* Active labor (regular contraction and> 4cm cervical opening)
* Placental anomaly
* Previous uterine surgery
* Chorioamnionitis
* Premature rupture of membranes
* Additional disease will affect tissue healing
* Body mass index BMI> 35kg / m2
* Consuming tobacco and / or alcohol
* Needing blood transfusion
* Multiple pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Since this is a study done at the time of cesarean section, only females are eligible.
Enrollment: 80 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Presence of isthmocele | 3 months
  The presence of an isthmocele (minimum 2 mm x 2 mm) identified on a transvaginal ultrasound 3 months after the cesarean section
Measurement of residual myometrial thickness | 3 months
  Measurement of residual myometrial thickness on a transvaginal ultrasound 3 months after the cesarean section

SECONDARY OUTCOMES:
Additional hemostatic sutures | Through the surgery completion, an average of 30 minutes
  Number of additional hemostatic sutures placed in the uterus
Operation time | Through the surgery completion, an average of 30 minutes
  Length of surgery from skin to delivery and delivery to skin closure (minutes)
Changes in Hemoglobin | 24 hours
  Changes in Hemoglobin from pre-operative measurement to post-operative measurement
Measurement of uterus | 3 months
  Measurements of uterus on a transvaginal ultrasound 3 months after the cesarean section( Uterus Length, Uterine position, Isthmocele depth, Isthmocele width, Cervical thickness, Fundus isthmocele distance, Isthmocele cervix distance, Hypoechoic isthmocele width in transverse plane)

CONTACTS AND LOCATIONS:
Overall Officials: Ilhan B Delibasi, A. Prof., Principal Investigator — Gaziosmanpasa University Obstetrics and Gynecology department; Kaan E Uzun, M.D., Study Chair — Gaziosmanpasa University Obstetrics and Gynecology department
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: No end date.
Access Criteria: Anyone who wishes to access the data. Any purpose. Data was saved on Mendeley data but it will be published after the article publication.